CLINICAL TRIAL: NCT05554783
Title: Analysis of Passive Leg Raise Test on Blood Pressure in Critically Ill Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: PLRonBP
Record Dates: First submitted 2022-04-21; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Shock; Hypovolemia; Hemodynamic Instability
MeSH Terms: conditions — Shock; Hypovolemia | interventions — Head-Down Tilt

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Trendelenburg position — Positioning the patient with head 15 degrees down

SUMMARY:
Positioning intensive care patients in Trendelenburg position to identify fluid responsiveness assessed by PiCCO device.

DETAILED DESCRIPTION:
It is a prospective observational study. Patients admitted to Intensive Care Unit of University Clinical Centre of Gdańsk, receiving advanced hemodynamic monitoring with PiCCO method will be enrolled. After blood pressure measurement, PiCCO will be calibrated with transpulmonary thermodilution with 10 - 20 ml of cold saline. Readings will be noted. The patient will be positioned in Trendelenburg position with it's head 15 degrees down. The increase of blood pressure after positioning in relation to the values obtained before the trial will be correlated to the parameters that asses patent's volaemia. After 5 minutes patient will be back to supine position and hemodynamic parameters will be recorded for another 5 minute.

ELIGIBILITY:
Inclusion Criteria:

* hemodynamic instability
* mechanical ventilation

Exclusion Criteria:

* increased intracranial pressure
* increased intraabdominal pressure
* lower limbs sequential compression system
* agitation
* patients exposed to pain stimulus before the test
* aortic aneurysm
* left to right cardiac shunt
* severe valvular insufficiency

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Intensive Care Unit of University Clinical Centre in Gdańsk
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of SVV with increase in blood pressure | 10 minutes
  Stroke volume variation (SVV) is a validated parameter that assess fluid responsiveness. In patients in whom SVV value is higher, theoretically Trendelenburg position will increase blood pressure in greater degree, than in patients in whom SVV is lower. We want to identify whether such correlation exist.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stefaniak, M.D., Principal Investigator — Medical University of Gdańsk, Department of Anesthesiology and Intensive Therapy; Radosław Owczuk, M.D., Ph.D., Study Director — Medical University of Gdańsk, Department of Anesthesiology and Intensive Therapy
Locations (1):
- Medical University of Gdańsk - Department of Anesthesiology and Intensive Care, Gdansk, Pomeranian Voivodeship, Poland